CLINICAL TRIAL: NCT05878106
Title: Creatine Supplementation and Resistance Training in Patients With Breast Cancer (CaRTiC Study)
Brief Title: Creatine Supplementation and Resistance Training in Patients With Breast Cancer
Acronym: CaRTiC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Collaborators: Hospital de Cruces (Other); Hospital de Basurto (Other); Poznan University of Medical Sciences (Other); Hospital Universitario de Burgos (Other); University of Calabria (Other)
Responsible Party: Principal Investigator, Arkaitz Castañeda, Principal Investigator, University of Deusto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CaRTiC
Record Dates: First submitted 2023-04-27; First posted 2023-05-26 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Supplementation; Resistance Training; Physical Performance; Quality of Life
MeSH Terms: conditions — Breast Neoplasms | interventions — Creatine; Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): They receive physical activity and nutrition recommendations.
- Resistance training group (Experimental): They will perform resistance training and placebo in the supplementation.
  Interventions: Other: Resistance training
- Resistance training and creatine supplementation group (Experimental): They will perform the same resistance training and will also receive creatine supplementation
  Interventions: Dietary Supplement: Creatine supplementation; Other: Resistance training

INTERVENTIONS:
Dietary Supplement: Creatine supplementation — 5 g/day supplementation of creatine for the duration of the exercise the 16-week intervention.
  The RG and the RCG will receive a supplement of soluble protein powder (20-30 g) daily.
  Arms: Resistance training and creatine supplementation group
Other: Resistance training — They will do resistance training. Resistance training will be a 16-week supervised workout that will consist of a series of resistance exercises (leg press, knee extension, knee bends, chest press, sit-ups, back extensions, pull-ups, and shoulder press) that involved the largest muscle groups of the body and will be performed three times a week on non-consecutive days.
  Arms: Resistance training and creatine supplementation group; Resistance training group

SUMMARY:
Background: Creatine supplementation is an effective ergogenic nutrient for athletes, as well as people for people starting a health or fitness program. Resistance training previously been identified as an important method of increasing muscle mass and strength among people, specially in people with cancer to avoid sarcopenia. The potential of creatine supplementation for adaptations produced by strength training in cancer patients are still unknown.

Objective: the primary aim of this study is to evaluate the effectiveness of a 16-week supervised resistance training program intervention with and without creatine supplementation in patients with breast cancer.

Methods: A multicentre, randomized, double-blind, placebo-controlled study designed to evaluate the effects of creatine supplementation in addition to resistance training in breast cancer patients. Patients will be randomly assigned to 3 groups: a control group (CG) and two experimental groups. The first resistance training group (RG) will perform resistance training, while the second resistance-creatine experimental group (RCG) will perform the same resistance training as the RG and will also receive a 5 g/day supplementation of creatine for the duration of the exercise the 16-week intervention. RG participants will follow the same daily dosing protocol, but in their case, with dextrose/maltodextrin. Resistance training will be a 16-week supervised workout that will consist of a series of resistance exercises (leg press, knee extension, knee bends, chest press, sit-ups, back extensions, pull-ups, and shoulder press) that involved the largest muscle groups of the body and will be performed three times a week on non-consecutive days. Both the RG and the RCG will receive a supplement of soluble protein powder (20-30 g) daily.

Discussion: The results of this intervention will help to better understand the potential of non-pharmacological treatment for improving strength and wellbeing values in breast cancer patients with and without creatine supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Stage pTis-T1-T2-T3 pN0-1 M0 (early stage).
* Patients who have completed local treatment [surgery + radiotherapy (RT)] undergoing clinical follow-up in outpatient clinics with or without adjuvant hormone therapy treatment.
* Age: ≥18-60 years.
* ECOG Performance status from 0 to 1 (IK ≥80%).
* Body mass index above than 18.5.
* Without excessive alcohol consumption (men > 21 and women > 14 units/week).
* No current or previous illness or injury that may prevent participation and training.
* No recent systematic strength training.
* Not taking medications that are known to alter body composition (corticosteroids, metformin...).
* People who carry out some aerobic training will not be excluded (the activity carried out will be recorded weekly).

Exclusion Criteria:

* Having received adjuvant or neoadjuvant chemotherapy.
* Metastatic carcinoma of the breast.
* Recurrence or second primary breast.
* History of previous cancer except previously treated basal cell carcinoma of the skin.
* Decompensated heart disease, uncontrolled hypertension (TAS>200 or TAD>110), heart failure (NYHA II or greater), heart failure or constrictive pericarditis, neutropenia, severe anemia (Hb<8.0 g/dl), blood count platelets <50,000 microL.
* Other health problems in which exercise is contraindicated
* Perform regular physical activity (150 min/week of moderate activity or 75 of vigorous activity), measured with the PVS questionnaire.
* Pregnancy.
* Criterion in the opinion of the investigator of inability to adequately understand the involvement and participation in this clinical study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Change in maximal resistance (upper and lower body) | 7 months follow up. Measures at 0, 2, 4 and 7 months.
  The maximal resistance in the upper and lower body will be measured in terms of the 5-repetition maximum test (5RM) (i.e. the maximum load that can be lifted five times) in chest and leg press exercises, respectively. Also a handgrip dynamometry test will be used to measure grip resistance.
Genetic study | Month 0
  Saliva samples will be taken from the participants using buccal swabs (4N6FLOQSwab, Life Technologies, Carlsbad, CA). The genetic analysis will be performed using Biomark HD system microfluidic analysis technology (Fluidigm, South San Francisco, CA). From that analysis DNA will be extracted using the QIAmp DNA Mini kit (Qiagen, Hilden, Germany) and will be quantified fluorometrically using Qubit (LifeTechnologies).
Change in Micro RNA (mRNA) | Month 0 and 4
  A 5/10 ml of urine will be collected in a 15 ml sterile plastic universal container tube kept at room temperature no more than 60 minutes, then stored at -20°C. Total RNA will be extracted from 400 μl of urine by using miRNeasy Serum/Plasma Kit (QIAGEN).

SECONDARY OUTCOMES:
Change in Physical function (walking) | 7 months follow up. Measures at 0, 2, 4 and 7 months.
  Physical function is assessed by the 6 Minute Walk Test (6MWT) in a 20-meter corridor. Is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Change in Physical function (sitting) | 7 months follow up. Measures at 0, 2, 4 and 7 months.
  A 30-s chair test will be performed performed to measure functional capacity. The number of stands a person can complete in 30 seconds will be recorded.
Change in Body composition | 7 months follow up. Measures at 0, 2, 4 and 7 months.
  Body composition (percentages of type of tissue) will be measured using a bioelectrical impedance analysis (Inbody 770, In-Bldg).
Change in dietary pattern | 7 months follow up. Measures at 0, 2, 4 and 7 months.
  Habitual food consumption and nutrient intake will be evaluated using the dietary history questionnaire.
Change in Gastrointestinal discomfort | 7 months follow up. Measures at 0, 2, 4 and 7 months.
  The unidimensional Gastrointestinal Function questionnaire was used to assess gastrointestinal discomfort. This questionnaire consists of 9 items with a frequency scale of 4 response options [none (0 points), mild (1 point), moderate (2 points) and severe (3 points)].
Change in Quality of life (general) | 7 months follow up. Measures at 0, 2, 4 and 7 months.
  The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) is used to assess general health-related quality of life status across physical functioning, physical role functioning, bodily pain, general health, vitality, social functioning, emotional role functioning, and mental health domains (higher scores indicating a greater quality of life). with scores for each of these scales (or dimensions) ranging from 0 to 100. Higher scores indicate higher quality of life.
Change in Quality of life (cancer specific) | 7 months follow up. Measures at 0, 2, 4 and 7 months.
  Cancer-specific quality of life is evaluated by the core quality of life (QLQ-C-30) questionnaire developed by the European Organization for Research and Treatment of Cancer (EORTC). This questionnaire includes five functional domains (physical, role, cognitive, emotional, and social, with higher scores representing greater function/quality of life) and three symptom scales (fatigue, pain, and nausea, with lower scores indicating greater quality of life/less symptom severity).
Change in fatigue level | 7 months follow up. Measures at 0, 2, 4 and 7 months.
  The cancer-related fatigue is assessed using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) scale. For all FACIT scales and symptom indices, the higher the score the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Arkaitz Castañeda, PhD, Principal Investigator — University of Deusto
Locations (1):
- Hospital de Cruces, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boidin M, Dawson EA, Thijssen DHJ, Erskine RM. VEGFA rs2010963 GG genotype is associated with superior adaptations to resistance versus endurance training in the same group of healthy, young men. Mol Genet Genomics. 2023 Jan;298(1):119-129. doi: 10.1007/s00438-022-01965-4. Epub 2022 Nov 3. PMID 36326960
- [Background] Brosnan ME, Brosnan JT. The role of dietary creatine. Amino Acids. 2016 Aug;48(8):1785-91. doi: 10.1007/s00726-016-2188-1. Epub 2016 Feb 13. PMID 26874700
- [Background] Buford TW, Kreider RB, Stout JR, Greenwood M, Campbell B, Spano M, Ziegenfuss T, Lopez H, Landis J, Antonio J. International Society of Sports Nutrition position stand: creatine supplementation and exercise. J Int Soc Sports Nutr. 2007 Aug 30;4:6. doi: 10.1186/1550-2783-4-6. No abstract available. PMID 17908288
- [Background] Campos-Ferraz PL, Gualano B, das Neves W, Andrade IT, Hangai I, Pereira RT, Bezerra RN, Deminice R, Seelaender M, Lancha AH. Exploratory studies of the potential anti-cancer effects of creatine. Amino Acids. 2016 Aug;48(8):1993-2001. doi: 10.1007/s00726-016-2180-9. Epub 2016 Feb 12. PMID 26872655
- [Background] Candow DG, Forbes SC, Chilibeck PD, Cornish SM, Antonio J, Kreider RB. Effectiveness of Creatine Supplementation on Aging Muscle and Bone: Focus on Falls Prevention and Inflammation. J Clin Med. 2019 Apr 11;8(4):488. doi: 10.3390/jcm8040488. PMID 30978926
- [Background] Chen JF, Tao Y, Li J, Deng Z, Yan Z, Xiao X, Wang DZ. microRNA-1 and microRNA-206 regulate skeletal muscle satellite cell proliferation and differentiation by repressing Pax7. J Cell Biol. 2010 Sep 6;190(5):867-79. doi: 10.1083/jcb.200911036. PMID 20819939
- [Background] Cornelissen VA, Defoor JG, Stevens A, Schepers D, Hespel P, Decramer M, Mortelmans L, Dobbels F, Vanhaecke J, Fagard RH, Vanhees L. Effect of creatine supplementation as a potential adjuvant therapy to exercise training in cardiac patients: a randomized controlled trial. Clin Rehabil. 2010 Nov;24(11):988-99. doi: 10.1177/0269215510367995. Epub 2010 Jun 24. PMID 20576665
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Dolan E, Artioli GG, Pereira RMR, Gualano B. Muscular Atrophy and Sarcopenia in the Elderly: Is There a Role for Creatine Supplementation? Biomolecules. 2019 Oct 23;9(11):642. doi: 10.3390/biom9110642. PMID 31652853
- [Background] Erskine RM, Williams AG, Jones DA, Stewart CE, Degens H. The individual and combined influence of ACE and ACTN3 genotypes on muscle phenotypes before and after strength training. Scand J Med Sci Sports. 2014 Aug;24(4):642-8. doi: 10.1111/sms.12055. Epub 2013 Feb 5. PMID 23384112
- [Background] Fairman CM, Kendall KL, Newton RU, Hart NH, Taaffe DR, Chee R, Tang CI, Galvao DA. Examining the effects of creatine supplementation in augmenting adaptations to resistance training in patients with prostate cancer undergoing androgen deprivation therapy: a randomised, double-blind, placebo-controlled trial. BMJ Open. 2019 Sep 20;9(9):e030080. doi: 10.1136/bmjopen-2019-030080. PMID 31542747
- [Background] Fenech M, El-Sohemy A, Cahill L, Ferguson LR, French TA, Tai ES, Milner J, Koh WP, Xie L, Zucker M, Buckley M, Cosgrove L, Lockett T, Fung KY, Head R. Nutrigenetics and nutrigenomics: viewpoints on the current status and applications in nutrition research and practice. J Nutrigenet Nutrigenomics. 2011;4(2):69-89. doi: 10.1159/000327772. Epub 2011 May 28. PMID 21625170
- [Background] Gerland L, Baumann FT, Niels T. Resistance Exercise for Breast Cancer Patients? Evidence from the Last Decade. Breast Care (Basel). 2021 Dec;16(6):657-663. doi: 10.1159/000513129. Epub 2021 Jan 28. PMID 35087367
- [Background] Giallauria F, Cittadini A, Smart NA, Vigorito C. Resistance training and sarcopenia. Monaldi Arch Chest Dis. 2016 Jun 22;84(1-2):738. doi: 10.4081/monaldi.2015.738. PMID 27374049
- [Background] Hall M, Trojian TH. Creatine supplementation. Curr Sports Med Rep. 2013 Jul-Aug;12(4):240-4. doi: 10.1249/JSR.0b013e31829cdff2. PMID 23851411
- [Background] Hardee JP, Porter RR, Sui X, Archer E, Lee IM, Lavie CJ, Blair SN. The effect of resistance exercise on all-cause mortality in cancer survivors. Mayo Clin Proc. 2014 Aug;89(8):1108-15. doi: 10.1016/j.mayocp.2014.03.018. Epub 2014 Jun 21. PMID 24958698
- [Background] Iannone F, Montesanto A, Cione E, Crocco P, Caroleo MC, Dato S, Rose G, Passarino G. Expression Patterns of Muscle-Specific miR-133b and miR-206 Correlate with Nutritional Status and Sarcopenia. Nutrients. 2020 Jan 22;12(2):297. doi: 10.3390/nu12020297. PMID 31979011
- [Background] Kim HJ, Kim CK, Carpentier A, Poortmans JR. Studies on the safety of creatine supplementation. Amino Acids. 2011 May;40(5):1409-18. doi: 10.1007/s00726-011-0878-2. Epub 2011 Mar 12. PMID 21399917
- [Background] Kreider RB, Kalman DS, Antonio J, Ziegenfuss TN, Wildman R, Collins R, Candow DG, Kleiner SM, Almada AL, Lopez HL. International Society of Sports Nutrition position stand: safety and efficacy of creatine supplementation in exercise, sport, and medicine. J Int Soc Sports Nutr. 2017 Jun 13;14:18. doi: 10.1186/s12970-017-0173-z. eCollection 2017. PMID 28615996
- [Background] Kreider RB, Stout JR. Creatine in Health and Disease. Nutrients. 2021 Jan 29;13(2):447. doi: 10.3390/nu13020447. PMID 33572884
- [Background] Lonbro S, Dalgas U, Primdahl H, Overgaard J, Overgaard K. Feasibility and efficacy of progressive resistance training and dietary supplements in radiotherapy treated head and neck cancer patients--the DAHANCA 25A study. Acta Oncol. 2013 Feb;52(2):310-8. doi: 10.3109/0284186X.2012.741325. Epub 2012 Nov 28. PMID 23190359
- [Background] Chandrashekhar Iyer L, Vaishali K, Babu AS. Prevalence of sarcopenia in heart failure: A systematic review. Indian Heart J. 2023 Jan-Feb;75(1):36-42. doi: 10.1016/j.ihj.2022.12.004. Epub 2022 Dec 22. PMID 36567064
- [Background] Norman K, Stubler D, Baier P, Schutz T, Ocran K, Holm E, Lochs H, Pirlich M. Effects of creatine supplementation on nutritional status, muscle function and quality of life in patients with colorectal cancer--a double blind randomised controlled trial. Clin Nutr. 2006 Aug;25(4):596-605. doi: 10.1016/j.clnu.2006.01.014. Epub 2006 May 15. PMID 16701923
- [Background] Padilha CS, Marinello PC, Galvao DA, Newton RU, Borges FH, Frajacomo F, Deminice R. Evaluation of resistance training to improve muscular strength and body composition in cancer patients undergoing neoadjuvant and adjuvant therapy: a meta-analysis. J Cancer Surviv. 2017 Jun;11(3):339-349. doi: 10.1007/s11764-016-0592-x. Epub 2017 Jan 4. PMID 28054255
- [Background] Patra S, Ghosh A, Roy SS, Bera S, Das M, Talukdar D, Ray S, Wallimann T, Ray M. A short review on creatine-creatine kinase system in relation to cancer and some experimental results on creatine as adjuvant in cancer therapy. Amino Acids. 2012 Jun;42(6):2319-30. doi: 10.1007/s00726-011-0974-3. Epub 2011 Jul 19. PMID 21769499
- [Background] Pescatello LS, Kostek MA, Gordish-Dressman H, Thompson PD, Seip RL, Price TB, Angelopoulos TJ, Clarkson PM, Gordon PM, Moyna NM, Visich PS, Zoeller RF, Devaney JM, Hoffman EP. ACE ID genotype and the muscle strength and size response to unilateral resistance training. Med Sci Sports Exerc. 2006 Jun;38(6):1074-81. doi: 10.1249/01.mss.0000222835.28273.80. PMID 16775548
- [Background] Soares RJ, Cagnin S, Chemello F, Silvestrin M, Musaro A, De Pitta C, Lanfranchi G, Sandri M. Involvement of microRNAs in the regulation of muscle wasting during catabolic conditions. J Biol Chem. 2014 Aug 8;289(32):21909-25. doi: 10.1074/jbc.M114.561845. Epub 2014 Jun 2. PMID 24891504
- [Background] Stares A, Bains M. The Additive Effects of Creatine Supplementation and Exercise Training in an Aging Population: A Systematic Review of Randomized Controlled Trials. J Geriatr Phys Ther. 2020 Apr/Jun;43(2):99-112. doi: 10.1519/JPT.0000000000000222. PMID 30762623
- [Background] Zhang G, Li X, Sui C, Zhao H, Zhao J, Hou Y, DU Y. Incidence and risk factor analysis for sarcopenia in patients with cancer. Oncol Lett. 2016 Feb;11(2):1230-1234. doi: 10.3892/ol.2015.4019. Epub 2015 Dec 9. PMID 26893724
- [Background] Pinheiro PA, Carneiro JA, Coqueiro RS, Pereira R, Fernandes MH. "Chair Stand Test" as Simple Tool for Sarcopenia Screening in Elderly Women. J Nutr Health Aging. 2016 Jan;20(1):56-9. doi: 10.1007/s12603-016-0676-3. PMID 26728934
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Cella D, Nowinski CJ. Measuring quality of life in chronic illness: the functional assessment of chronic illness therapy measurement system. Arch Phys Med Rehabil. 2002 Dec;83(12 Suppl 2):S10-7. doi: 10.1053/apmr.2002.36959. PMID 12474167